CLINICAL TRIAL: NCT02973867
Title: Myokines Role in Bone Mineral Density Increase During Obesity
Brief Title: Myokines Role During Obesity
Acronym: Bonamy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9768
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Obesity, Adolescent
Keywords: Bone mineral density; Myokines; Adipokines
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort called Elodie: Obese patients

SUMMARY:
We showed, for the first time, that Z-score increase during obesity was dependent on sex, severity of obesity and age but also on the bone site. Although the increase in BMD at bearing areas seems to be logically explained by the assumption that mechanical stresses have an osteogenic effect on bone tissue, BMD can in no way respond to the concomitant increase in BMD at non-load bearing areas such as the radius. These results suggest that changes in certain systemic compounds, induced by obesity, may interfere with bone metabolism. Moreover, the fact that the BMD or Z score is positively and only correlated with muscle mass and not with fat mass confirm that mechanical stresses are not the only factors acting on bone tissue.

Our objectives are to determine the relationship between plasma concentration of myokines, adipokines, bone markers and BMD in obese subjects.

DETAILED DESCRIPTION:
We showed, for the first time, that Z-score increase during obesity was dependent on sex, severity of obesity and age but also on the bone site. Although the increase in BMD at bearing areas seems to be logically explained by the assumption that mechanical stresses have an osteogenic effect on bone tissue, BMD can in no way respond to the concomitant increase in BMD at non-load bearing areas such as the radius. (Maïmoun L and Col Bone 2015 Dec 1. S8756-3282 (15) 00421-4). These results suggest that changes in certain systemic compounds, induced by obesity, may interfere with bone metabolism. Moreover, the fact that the BMD or Z score is positively and only correlated with muscle mass and not with fat mass confirm that mechanical stresses are not the only factors acting on bone tissue.

Our objectives are to determine the relationship between plasma concentration of myokines, adipokines, bone markers and BMD in obese subjects.

Our objectives are to determine the relationship between plasma concentration of myokines (myostatin, follistatin), adipokines (leptin, adiponectin) and bone markers (CTX, Trap5, P1NP, ostéocalcin) in a cohort of obese patients, with differents obesity severity, differents ages.

ELIGIBILITY:
Inclusion Criteria:

* obese patients age above 18 years old

Exclusion Criteria:

* non agreement of inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
myosin concentration | 1 day
  blood measure

SECONDARY OUTCOMES:
adipokines concentration | 1 day
  blood measure

CONTACTS AND LOCATIONS:
Overall Officials: SULTAN ARIANE, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided